CLINICAL TRIAL: NCT04803500
Title: Restoration of Immediate Peri-implant Defect by Simvastatin: a Controlled Clinical and Cone Beam Computed Tomography Study
Brief Title: Simvastatin Around Immediate Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mina Adel Rizk Botros, Assistant Researcher, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PER 15-1M
Record Dates: First submitted 2021-02-07; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Immediate Implant Placement; Bone Regeneration; Alveolar Bone Resorption
Keywords: Simvastatin; Immediate implant placement; gap distance; ridge dimension alteration; cone beam computed tomopgraphy
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin group (Active Comparator): simvastatin gel (1.2 mg/0.1 ml of solid lipid nanoparticles) was locally applied to fill the jumping distance.
  Interventions: Drug: Simvastatin
- Control group (Placebo Comparator): the solid lipid nanoparticles carrier was injected into the jumping distance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — single injection of simvastatin gel in the gap around immediately placed implant
  Arms: Simvastatin group
Drug: Placebo — single injection of the solid lipid nanoparticle carrier in the gap around immediately placed implant
  Arms: Control group

SUMMARY:
The study evaluated the effect of local application of simvastatin around immediate implant on the amount of gap fill, ridge dimensional alterations and bone density in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 50 years old
* requiring the extraction of 2 non-restorable maxillary canine or premolar on each side of the arch
* following extraction, the crestal bone had to be located 3 mm apical to the free gingival margin
* at least 3 mm of bone beyond the root apex was required to guarantee implant primary stability

Exclusion Criteria:

* unstable systemic diseases precluding surgical procedures
* compromised general health conditions that would impair bone healing including present history of bone irradiation, patient on bisphosphonates therapy, antitumor chemotherapy
* pregnancy
* compromised healing conditions e.g. uncontrolled diabetes mellitus

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-05-03 (Actual)

PRIMARY OUTCOMES:
Effect of simvastatin on gap fill | 3 months after implant placement
  using cone beam computed tomography
Effect of simvastatin on horizontal ridge dimension | 3 months after implant placement
  using cone beam computed tomography
Effect of simvastatin on crestal bone level | 3 months after implant placement
  using cone beam computed tomography
Effect of simvastatin on bone density | 3 months after implant placement
  using cone beam computed tomography

SECONDARY OUTCOMES:
Quality of wound healing | 1 week after implant placement
  wound healing index
Quality of wound healing | 2 weeks after implant placement
  wound healing index

IPD SHARING:
Plan to Share IPD: Yes